CLINICAL TRIAL: NCT00613977
Title: Pilot Study-A Cost and Time Savings Comparison of Lamellar Body Count and FLM II
Brief Title: Comparison of Two Fetal Lung Maturity Tests
Status: Withdrawn | Type: Observational
Why Stopped: Withdrawn
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 2007013
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Respiratory Distress Syndrome
Keywords: fetal lung maturity; lamellar body count
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Amniotic fluid for fetal lung maturity test
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators wish to compare the difference in both cost and time to result for determining fetal lung maturity for the Lamellar Body Count method and the Fetal Lung Maturity II. Our hypothesis is that the time to result will be significantly less using the Lamellar Body Count method, and the cost associated with this method over the traditional FLM II will be favorable.

DETAILED DESCRIPTION:
Rationale/Background: This pilot study is a prospective cohort analysis of two methods currently available at our institution for the determination of fetal lung maturity (FLM) using amniotic fluid. The investigators wish to explore a cost and time savings potential between these two available tests. The test most utilized for the determination of FLM is the evaluation of phospholipids from the amniotic fluid. In our particular institution, the relationship of surfactant to albumin (S/A ratio) is analyzed using a measured fluorescent polarization called the FLM II procedure performed on the TDx or TDxFLx chemical analyzer which is commercially available from Abbott Labs. This test is time-consuming and not available at all institutions.

Lamellar bodies are lamellated phospholipids that represent a storage form of surfactant (1). Because lamellar body diameter (range, 1-5 µm) is similar to that of small platelets, lamellar body counts (LBCs) can be obtained rapidly with use of the platelet channel of a hematology analyzer. The investigators wish to compare the difference in both cost and time to result for determining FLM for the LBC method and the FLM II. Our hypothesis is that the time to result will be significantly less using the LBC method, and the cost associated with this method over the traditional FLM II will be favorable.

Extensive research has shown the efficacy of analyzing fetal lung maturity using lamellar bodies (2-11). Since the efficacy of this method has been established, the adequacy of the lamellar body count in comparison to the FLM II is not in question in this study. While other studies have speculated that a cost and time savings would exist, no literature was found to answer this precise question. The authors feel this information could benefit the medical community from an economic standpoint.

Amniotic fluid collected at the time of amniotomy on term cesarean sections will be sent to OSUMC laboratory for FLM analysis using both a LBC and the FLM II. Our hypothesis is that both the time to result and cost using the LBC method will be substantially less.

Methodology Mechanism of Testing At present, FLM testing at Oklahoma State University Medical Center (OSUMC) is performed by TDx-FLM chemical analyzer manufactured by Abbott Labs. Most laboratories using the Abbott FLM-II assay for assessing fetal lung maturity follow the manufacturer's recommendations for interpreting the surfactant to albumin ratio. Thus, values greater than 55 mg/g are considered mature and values less than 40 mg/g immature. McElrath et al., reported a probability of respiratory distress syndrome (RDS) of 15% or less can be achieved with a S/A ratio cutoff of 60 mg or more at 28 weeks of gestation, 50 or more at 30 weeks, 40 or more at 33 weeks, 30 or more at 35 weeks, and 20 or more at 37 weeks (12).

Lamellar bodies have been tested on many hospital instruments that are used for the hematology testing at their institutions. The ADVIA 2120 (Siemens Medical Solutions Diagnostics, Tarrytown, NY), which is a flow cytometry system that functions to identify and count specific cells in body fluid, is used in the OSUMC laboratory for hematology and other body fluids. Although it has not been used for LBC in our institution, it certainly has that capability according to the manufacturer (13). Neerhof et. al, recently described a change in the threshold at their particular institution. The level of maturity was increased from 30,000 to 50,000 LB/ul. This resulted in significantly fewer neonatal intensive care unit admissions for RDS (14).

An algorithm to FLM testing first utilizing the LBC has been published by Ventolini et al. This algorithm is pictured in Figure 1 (15). We will incorporate this algorithm into our cost analysis as indeterminate LBC values would have required the FLM II procedure, thus elevating the cost for that patient.

Amniotic fluid will be obtained by the operating surgeon or assistant once amniotomy is made. At least 2 ml of amniotic fluid is required for both tests. The fluid will them be handed off to waiting nursing personnel. Once the amniotic fluid is obtained, LBC and S/A ratios will be sent to the laboratory as a stat order. Laboratory personnel will record the time that the specimen is checked into lab and the time the result is available, which is their standard protocol. These times will be used to calculate the time differences between LBC and S/A ratios. The patient will be identified by their assigned medical record number in the hospital. Details of the LBC protocol using the ADVIA 2120 can be found in Table 1.

We will record results of both studies. When an indeterminate level is obtained using the lamellar body count, a cost for performing the FLM II procedure will be added to the lamellar body count cost for that particular patient. The amount that would have been charged to the patient will be used to calculate the cost savings in our sample size. We will then compare the cost of the LBC, LBC and TDxFLM (if required by our algorithm), and the TDxFLM alone.

Study Population:

The study population will include ten term gestations scheduled for either repeat cesarean section (C/S) or primary C/S for malpresentation. Term will be defined as 37 completed weeks based on a sure last menstrual period or first trimester ultrasound crown rump length measurement.

Consent will be obtained either in the resident clinic or on the morning of the scheduled procedure. The resident investigator or one of the obstetrical residents at OSUMC will consent the patient.. The residents participating in consenting will be given instructions regarding the consent process as well as inclusion/exclusion criteria.

The cost for both laboratory tests will be approximately $45 per patient. The sample size will be limited by a research grant of $500.00 provided by the Osteopathic Founders Foundation. Other funding is in application and expansion of this project will be likely in the future.

Inclusion Criteria:

* Term intrauterine gestations beyond 37 completed weeks with dating calculated by their sure last menstrual period (LMP) using Negel's rule or utilizing a first trimester crown rump length ultrasound.
* Women with a previous C/S scheduled for repeat C/S.
* Women who are undergoing a scheduled C-Section for malpresentation

Exclusion Criteria:

* Presence of gross blood in amniotic sample
* Hematocrit count greater than 1% on ADVIA 2120
* Presence of meconium in sample
* Patients with oligohydramnios defined as an amniotic fluid index of less than 5 cm or polyhydramnios defined as an amniotic fluid index of more than 24 cm.

Early Termination Criteria:

If for any reason the investigators or the obstetrician performing the C/S believe the patient or fetus may be harmed by the extra time required for amniotic fluid collection (albeit short), the patient may be removed from the study without her consent. The volunteer would also have the right to terminate her participation in the study and to terminate the investigators' rights to use the collected fluid or analyzed result at any time.

Collection Sheet Appendix C "Lamellar Body Data Collection Sheet" will be used for the collection and storage of data. All information will be de-identified for the collection, storage and retrieval of information.

Data Collection Only the principle investigator(s) will have access to the patients' data collection sheet. Individual physicians involved in the care of a specific patient will have access to that patient's information. All individuals will be in compliance with HIPPA guidelines as set forth by the university and the medical center. Treatment decisions will not be based on the results of data collected for this study.

The following information will be obtained from the patients chart for entry on the data collection sheet.

1. Maternal age
2. Gravity/Parity
3. Estimated Gestational Age and how that was figured
4. Maternal complications - diabetes, hypertension, PIH, coronary vascular disease, thyroid disease, thrombophilia,
5. Date collected
6. Time collected
7. Time received
8. Time reported - FLM, LB
9. Difference in total times
10. FLM result - mature, intermediate or immature
11. LB result - mature, intermediate or immature
12. Cost for FLM
13. Cost for LB No other data will be collected from any patient charts. The resident investigator will assist in the collection of data and will have qualifications for basic human research and HIPPA training as they fall under the OSU - CHS community of individuals with this privilege. Further, physicians and residents which have direct access to current patients chart in their medical management will determine needs for fluid collections and assist in patient consents.

Analysis: An algebraic expression will be used to determine which procedure is the most time and cost effective. Let P be the proportion of LBC's that have conclusive results. Let X denote an attribute of LBC (say cost or time) and let Y denote the same attribute for FLM II. The following equation asks the question "when are the costs associated with just performing FLM II greater than the costs associated with LBC with the FLM II backup?"

Cost (or time) of LBC with FLM II back up < Cost (or time) of FLM II

when

X < P*Y

In other words: Using LBC is beneficial when the proportion of conclusive results is greater than the proportion of cost of LBC over FLM II.

Confidentiality: All records and lab results will be maintained at Oklahoma State University Medical Center, department of medical records and laboratory storage on the hospital's Meditech system. Research analysis data collection sheets will be de-identified and will be maintained by the Department of Ob/Gyn in a secured location at 717 South Houston Ave, Tulsa OK 74127.

ELIGIBILITY:
Inclusion Criteria:

* Term intrauterine gestations beyond 37 completed weeks with dating calculated by their sure last menstrual period (LMP) using Negel's rule or utilizing a first trimester crown rump length ultrasound.
* Women with a previous C/S scheduled for repeat C/S.
* Women who are undergoing a scheduled C-Section for malpresentation

Exclusion Criteria:

* Presence of gross blood in amniotic sample
* Hematocrit count greater than 1% on ADVIA 2120
* Presence of meconium in sample
* Patients with oligohydramnios defined as an amniotic fluid index of less than 5 cm or polyhydramnios defined as an amniotic fluid index of more than 24 cm.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women delivering a term infant by cesarean section at Oklahoma State University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
cost/time to run test | six months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Johnson, D.O., Principal Investigator — OSU Center for Health Sciences Dept of Ob/Gyn
Locations (1):
- Oklahoma State University Medical Center, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Weaver TE, Na CL, Stahlman M. Biogenesis of lamellar bodies, lysosome-related organelles involved in storage and secretion of pulmonary surfactant. Semin Cell Dev Biol. 2002 Aug;13(4):263-70. doi: 10.1016/s1084952102000551. PMID 12243725
- [Background] Fakhoury G, Daikoku NH, Benser J, Dubin NH. Lamellar body concentrations and the prediction of fetal pulmonary maturity. Am J Obstet Gynecol. 1994 Jan;170(1 Pt 1):72-6. doi: 10.1016/s0002-9378(94)70386-8. PMID 8296848
- [Background] Pearlman ES, Baiocchi JM, Lease JA, Gilbert J, Cooper JH. Utility of a rapid lamellar body count in the assessment of fetal maturity. Am J Clin Pathol. 1991 Jun;95(6):778-80. doi: 10.1093/ajcp/95.6.778. PMID 2042585
- [Background] Bowie LJ, Shammo J, Dohnal JC, Farrell E, Vye MV. Lamellar body number density and the prediction of respiratory distress. Am J Clin Pathol. 1991 Jun;95(6):781-6. doi: 10.1093/ajcp/95.6.781. PMID 2042586
- [Background] Ashwood ER, Palmer SE, Taylor JS, Pingree SS. Lamellar body counts for rapid fetal lung maturity testing. Obstet Gynecol. 1993 Apr;81(4):619-24. PMID 8459979
- [Background] Dalence CR, Bowie LJ, Dohnal JC, Farrell EE, Neerhof MG. Amniotic fluid lamellar body count: a rapid and reliable fetal lung maturity test. Obstet Gynecol. 1995 Aug;86(2):235-9. doi: 10.1016/0029-7844(95)00120-g. PMID 7617355
- [Background] Greenspoon JS, Rosen DJ, Roll K, Dubin SB. Evaluation of lamellar body number density as the initial assessment in a fetal lung maturity test cascade. J Reprod Med. 1995 Apr;40(4):260-6. PMID 7623354
- [Background] Lee IS, Cho YK, Kim A, Min WK, Kim KS, Mok JE. Lamellar body count in amniotic fluid as a rapid screening test for fetal lung maturity. J Perinatol. 1996 May-Jun;16(3 Pt 1):176-80. PMID 8817425
- [Background] Lewis PS, Lauria MR, Dzieczkowski J, Utter GO, Dombrowski MP. Amniotic fluid lamellar body count: cost-effective screening for fetal lung maturity. Obstet Gynecol. 1999 Mar;93(3):387-91. doi: 10.1016/s0029-7844(98)00416-5. PMID 10074985